CLINICAL TRIAL: NCT07392190
Title: A Phase 3 Randomized, Double-Blind, Placebo-Controlled Study to Investigate the Efficacy and Safety of Once Weekly Eloralintide in Adult Participants With Persistent Obesity or Overweight Treated With a Weekly Incretin, With and Without Type 2 Diabetes
Brief Title: A Study of Eloralintide (LY3841136) in Participants With Persistent Obesity Who Are Treated With a Weekly Incretin
Acronym: ENLIGHTEN-6
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 27743; J3R-MC-YDAL (Other: Eli Lilly and Company); 2025-523659-73-00 (EU CTIS Number)
Record Dates: First submitted 2026-01-30; First posted 2026-02-06 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Overweight; Obesity
Keywords: Amylin receptor agonist
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Eloralintide Dose 1 (Experimental): Participants will receive eloralintide subcutaneously (SC)
  Interventions: Drug: Eloralintide
- Eloralintide Dose 2 (Experimental): Participants will receive eloralintide SC
  Interventions: Drug: Eloralintide
- Eloralintide Dose 3 (Experimental): Participants will receive eloralintide SC
  Interventions: Drug: Eloralintide
- Eloralintide Dose 4 (Experimental): Participants will receive eloralintide SC
  Interventions: Drug: Eloralintide
- Placebo (Placebo Comparator): Participants will receive placebo SC
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Eloralintide — Administered SC
  Other Names: LY3841136
  Arms: Eloralintide Dose 1; Eloralintide Dose 2; Eloralintide Dose 3; Eloralintide Dose 4
Drug: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
The main purpose of this study is to evaluate the efficacy and safety of eloralintide compared with placebo in participants with persistent obesity or overweight, with or without type 2 diabetes, and on stable incretin background therapy.

Participation in the study will last about 80 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Are on stable incretin therapy at screening
* With persistent obesity or overweight defined as:

  * ≥30 kg/m2 OR
  * ≥27 kg/m2 with at least one existing obesity related complication at screening:

    * hypertension
    * dyslipidemia
    * obstructive sleep apnea
    * cardiovascular disease (for example, ischemic cardiovascular disease, New York Heart Association Functional Class I-III heart failure), or
    * type 2 diabetes
* Have a stable body weight (<5% body weight change) at screening

Exclusion Criteria:

* Have a prior or planned surgical treatment for obesity (liposuction, cryolipolysis, or abdominoplasty allowed if performed >1 year before screening)
* Have a prior or planned endoscopic procedure and/or device-based therapy for obesity (prior device-based therapy acceptable if device removal was more than 6 months prior to screening)
* Have type 1 diabetes
* Have taken any of the following antihyperglycemic medications within 90 days before screening:

  * dipeptidyl peptidase-4 (DPP-4) inhibitors
  * amylin analogs
  * insulin
* Have had within 90 days prior to screening:

  * heart attack
  * stroke
  * coronary artery revascularization
  * unstable angina, or
  * hospitalization due to congestive heart failure
* Have a history or diagnosis of New York Heart Association Functional Classification Class IV congestive heart failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2028-06 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Percent Change from Baseline in Body Weight | Baseline, Week 64

SECONDARY OUTCOMES:
Change from Baseline in Waist Circumference | Baseline, Week 64
Percent Change in Baseline in Triglycerides | Baseline, Week 64
Change from Baseline in Systolic Blood Pressure | Baseline, Week 64
Change from Baseline in Body Mass Index (BMI) | Baseline, Week 64
Change from Baseline in Fasting Glucose in Participants with Type 2 Diabetes at Baseline | Baseline, Week 64
Change from Baseline in Short Form-36 (SF-36 v2) Score | Baseline, Week 64
Change from Baseline in EQ-5D-5L Score | Baseline, Week 64
Change from Baseline in Control of Eating Questionnaire (CoEQ) Score | Baseline, Week 64
Achievement of Improved Categorical Shift in Patient Global Impression of Severity (PGIS) Physical Function Weight | Baseline, Week 64
Percent Change from Baseline in Fasting Insulin | Baseline, Week 64
Percent Change from Baseline in High Sensitivity C-Reactive Protein (hsCRP) | Baseline, Week 64
Change from Baseline in Estimated Glomerular Filtration Rate (eGFR) | Baseline, Week 64
Change in Medication Use | Baseline through Week 64
Pharmacokinetics (PK): Maximum Concentration at Steady State (Cmax,ss) | Baseline through Week 64
PK: Area Under the Concentration Versus Time Curve for One Dosing Interval at Steady State (AUC(0-ᴛ)ss) | Baseline through Week 64

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (178):
- United States (51):
  - Birmingham Clinical Research, Birmingham, Alabama
  - RIO Clinical Trials - Phoenix, Phoenix, Arizona
  - Headlands Research - Scottsdale, Scottsdale, Arizona
  - Novak Clinical Research - Tucson - North La Cholla Boulevard, Tucson, Arizona
  - Irvine Clinical Research, Irvine, California
  - Scripps Whittier Diabetes Institute, La Jolla, California
  - Peninsula Research Associates, Rolling Hills Estates, California
  - Care Access - Sacramento, Sacramento, California
  - Artemis Institute for Clinical Research, San Diego, California
  - Southern California Clinical Research, Santa Ana, California
  - University Clinical Investigators, Inc., Tustin, California
  - New England Research Associates, LLC, Bridgeport, Connecticut
  - Yale University School of Medicine, New Haven, Connecticut
  - Chase Medical Research, LLC, Waterbury, Connecticut
  - JEM Research Institute, Atlantis, Florida
  - AMR Clinical, Doral, Florida
  - Northeast Research Institute (NERI), Fleming Island, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - New Horizon Research Center, Miami, Florida
  - St Johns Center for Clinical Research, Saint Augustine, Florida
  - Metabolic Research Institute, Inc., West Palm Beach, Florida
  - Teak Research Consults - Dunwoody, Dunwoody, Georgia
  - Center for Advanced Research & Education, Gainesville, Georgia
  - Family First Medical Center, Idaho Falls, Idaho
  - Great Lakes Clinical Trials - Ravenswood, Chicago, Illinois
  - Iowa Diabetes and Endocrinology Research Center, West Des Moines, Iowa
  - Cotton O'Neil Diabetes & Endocrinology, Topeka, Kansas
  - AMR Clinical, Lexington, Kentucky
  - IMA Clinical Research Monroe - Armand, Monroe, Louisiana
  - Centennial Medical Group, Columbia, Maryland
  - Brigham and Women's Hospital Diabetes Program, Boston, Massachusetts
  - Great Lakes Research Institute, Southfield, Michigan
  - Arcturus Healthcare , PLC, Troy Internal Medicine Research Division, Troy, Michigan
  - Clinical Research Professionals, Chesterfield, Missouri
  - NYU Langone Health, New York, New York
  - Weill Cornell Medical College, New York, New York
  - IMA Clinical Research Manhattan, New York, New York
  - University of North Carolina Medical Center, Chapel Hill, North Carolina
  - Medication Management, Greensboro, North Carolina
  - Carteret Medical Group, Morehead City, North Carolina
  - Accellacare - Wilmington - 1917 Tradd Court, Wilmington, North Carolina
  - Care Access - Lima, Lima, Ohio
  - Preferred Primary Care Physicians, Preferred Clinical Research (Ofc 18), Pittsburgh, Pennsylvania
  - UT Southwestern Medical Center, Dallas, Texas
  - Juno Research, Houston, Texas
  - Synergy Groups Medical LLC - Missouri City, Missouri City, Texas
  - IMA Clinical Research San Antonio, San Antonio, Texas
  - Endeavor Clinical Trials, San Antonio, Texas
  - Consano Clinical Research, LLC, Shavano Park, Texas
  - Texas Valley Clinical Research, Weslaco, Texas
  - Medrasa Clinical Research, Wylie, Texas
- Australia (10):
  - Emeritus Research, Botany
  - Box Hill Hospital, Box Hill
  - Royal Brisbane and Women's Hospital, Brisbane
  - Emeritus Research, Camberwell
  - Barwon Health, Geelong
  - Austin Health - Repatriation Hospital, Heidelberg West
  - AIM Research, Merewether
  - Southern Adelaide Diabetes & Endocrine Services, Oaklands Park
  - Royal North Shore Hospital, St Leonards
  - Innovate Clinical Research, Waitara
- Belgium (9):
  - Imelda General Hospital, Bonheiden
  - Université Libre de Bruxelles - Hôpital Erasme, Brussels
  - Ziekenhuis Oost-Limburg, Campus St.-Jan, Genk
  - Jan Yperman Ziekenhuis, Ieper
  - AZ Groeninge Campus Kennedylaan, Kortrijk
  - UZ Leuven, Leuven
  - AZ Sint-Maarten, Mechelen
  - Meclinas, Mechelen
  - Az Damiaan vzw, Ostend
- Brazil (7):
  - Quanta Diagnóstico e Terapia, Curitiba
  - Centro de Diabetes Curitiba, Curitiba
  - Private Practice - Dr.Miguel N. Hissa, Fortaleza
  - CPCLIN, São Paulo
  - Hospital 9 De Julho, São Paulo
  - CEDOES, Vitória
  - Integral Pesquisa e Ensino, Votuporanga
- China (20):
  - Luhe Hospital, Beijing
  - The First Hospital of Jilin University, Changchun
  - The Second Hospital of Jilin University, Changchun
  - The Second Xiangya Hospital of Central South University, Changsha
  - Sichuan Provincial People's Hospital, Chengdu
  - West China Hospital Sichuan University, Chengdu
  - 2nd Affiliated Hospital Chongqing Medical Universi, Chongqing
  - Zhujiang Hospital, Guangzhou
  - The Affiliated Hospital of Guizhou Medical University, Guiyang
  - The Second People's Hospital of Hefei, Hefei
  - Huzhou Central Hospital, Huzhou
  - The First Affiliated Hospital of Henan University of Science &Technology, Luoyang Shi
  - Affiliated Hospital of Luzhou Medical College, Luzhou
  - Jiangxi Provincial People's Hospital, Nanchang
  - Nanjing First Hospital, Nanjing
  - Zhongda Hospital Southeast University, Nanjing
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjing
  - Ningbo First Hospital, Ningbo
  - Zhongshan Hospital,Fudan University, Shanghai
  - The Central Hospital of Wuhan, Wuhan
- Czechia (4):
  - Diahaza s.r.o., Holešov
  - MUDr. Michala Pelikanova s.r.o., Prague
  - Milan Kvapil s.r.o., Diabetologicka ambulance, Prague
  - ResTrial s.r.o., Prague
- India (12):
  - Motilal Nehru Medical College Hospital, Allahabād
  - Life Care Hospital and Research Centre, Bangalore
  - Madras Diabetes Research Foundation, Chennai
  - Nizam's Institute of Medical Sciences, Hyderabad
  - Eternal Heart Care Center and Research Institute, Jaipur
  - Atmaram Child Care, Kanpur
  - Shree Mahalaxmi DIATONE Institute, Kolhāpur
  - BSES MG Hospital, Mumbai
  - Mysore Medical College, Mysore
  - All India Institute of Medical Sciences (AIIMS) - Nagpur, Nagpur
  - Supe Heart & Diabetes Hospital and Research Centre, Nashik
  - Nirmal Hospital Pvt Ltd., Surat
- Israel (17):
  - Emek Medical Center, Afula
  - Clalit Health Services - Atlit, Atlit
  - Soroka Medical Center, Beersheba
  - Hillel Yaffe Medical Center, Hadera
  - Rambam Health Care Campus, Haifa
  - Edith Wolfson Medical Center, Holon
  - Hadassah Medical Center, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Maccabi health care services - Qiryat Motzkin, Kiryat Motzkin
  - Laniado Hospital, Netanya
  - Rabin Medical Center - Hasharon Campus, Petah Tikva
  - Rabin Medical Center, Petah Tikva
  - Sheba Medical Center, Ramat Gan
  - Kaplan Medical Center, Rehovot
  - Clalit Health Services - Sakhnin Community Clinic, Sakhnin
  - Diabetes Medical Center, Tel Aviv
  - Sourasky Medical Center, Tel Aviv
- Japan (11):
  - The Institute of Medical Science, Asahi Life Foundation, Chūōku
  - Rinku General Medical Center, Izumisano
  - Kanto Rosai Hospital, Kawasaki
  - Kimitsu Chuo Hospital, Kisarazu
  - Kure Medical Center, Kure
  - Takeda General Hospital - Kyoto, Kyoto
  - Mikannohana Clinic, Diabetes, Endocrinology and Metabolism, Matsuyama
  - Kansai Electric Power Hospital, Osaka
  - Manda Memorial Hospital, Sapporo
  - Shimonoseki Medical Center, Shimonoseki
  - Japanese Red Cross Society - Wakayama Medical Center, Wakayama
- Mexico (6):
  - Medical Center Metas, Chihuahua City
  - Private Practice - Dr. Arechavaleta Granell Maria del Rosario, Guadalajara
  - Invecordis S.C., Huixquilucan
  - Centro de Investigacion en Artritis y Osteoporosis SC, Mexicali
  - CEINV Salud, Monterrey
  - Clínica García Flores SC, Monterrey
- Puerto Rico (2):
  - Advanced Clinical Research, LLC, Bayamón
  - Isis Clinical Research Center, Guaynabo
- Romania (10):
  - Mariodiab Clinic, Brasov
  - C.M.D.T.A. Neomed, Brasov
  - Geea Medical Easy Diet, Bucharest
  - Centrul Medical NutriLife, Bucharest
  - Gama Diamed, Mangalia
  - Diabdana, Oradea
  - Clinica Korall, Satu Mare
  - Rinart Diab SRL, Târgovişte
  - SC Dentosim Queen SRL - Centrul Medical Diamed, Târgu Mureş
  - Cabinet Medical Dr.Geru, Timișoara
- Spain (10):
  - Hospital San Rafael - La Coruña, A Coruña
  - Centro Periférico de Especialidades Bola Azul, Almería
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Instituto Gallego de Cirugía Ocular, Ferrol
  - Clínica Juaneda, Palma de Mallorca
  - Hospital Universitario Quironsalud Madrid, Pozuelo de Alarcón
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Clínica nuevas Tecnologías en Diabetes y Endocrinología (NTDE), Seville
  - Hospital Quiron Infanta Luisa, Seville
  - Vithas Hospital Sevilla, Seville
- Taiwan (9):
  - Chiayi Christian Hospital, Chiayi City
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Chang Gung Memorial Hospital at Kaohsiung, Kaohsiung Niao Sung Dist
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Medical University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Medical Foundation-Linkou Branch, Taoyuan District

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication or approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/